CLINICAL TRIAL: NCT04145856
Title: Efficacy of the Combination Therapy With Alverine-simeticone and i3.1 Probiotic Formula in the Quality of Life of Patients With IBS-D or IBS-M in Hospital Juarez Mexico
Brief Title: Combination of Alverine-simeticone and i3.1 Probiotic in IBS-D and IBS-M in Mexico
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Juarez de Mexico (Other Government)
Responsible Party: Principal Investigator, Nuria Pérez López, Digestive Physiology Lab Head, Hospital Juarez de Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HJM 0492/18-R
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: Probiotic; Antispasmodic; Rome-IV
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Simethicone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): - Control arm
  Interventions: Other: Placebo
- Probiotic (Experimental): - Arm with active probiotic alone
  Interventions: Dietary Supplement: I31 probiotic
- Probiotic + Antispasmodic/Antifoam (Experimental): - Arm with active probiotic combined to antispasmodic/antifoam drug
  Interventions: Combination Product: I31 probiotic combined to Alverine/Simethicone

INTERVENTIONS:
Dietary Supplement: I31 probiotic — I31 probiotic formula (dietary supplement), consisting of 3 billion cfus of strains P. acidilactici CECT7483, L.plantarum CECT7484 and L.plantarum CECT7485, once daily (u.i.d)
  Arms: Probiotic
Combination Product: I31 probiotic combined to Alverine/Simethicone — * I31 probiotic formula (dietary supplement), consisting of 3 billion cfus of strains P. acidilactici CECT7483, L.plantarum CECT7484 and L.plantarum CECT7485, once daily (u.i.d)
  * Antispasmodic/antifoam drug, consisting of Alverine Citrate 60 mg and Simethicone 300 mg, thrice daily (t.i.d)
  Arms: Probiotic + Antispasmodic/Antifoam
Other: Placebo — Placebo treatment (maltodextrin), once daily (u.i.d)
  Arms: Placebo

SUMMARY:
This randomized study evaluates the usefulness of the I31 probiotic formula, alone or in combination with alverine/simethicone, against placebo, in the treatment of diarrhea-predominant or mixed irritable bowel syndrome

DETAILED DESCRIPTION:
Irritable Bowel Syndrome (IBS) is a functional gastrointestinal disease in which recurrent abdominal pain is associated with defecation or a change in bowel habits. Disordered bowel habits are typically present (ie, constipation, diarrhea, or a mix of constipation and diarrhea), as are symptoms of abdominal bloating/distention.

I31 is a probiotic formula composed of strains Pediococcus acidilactici CECT7483 and Lactobacillus plantarum CECT7484 and CECT7485, previously shown to improve quality of life in patients with IBS of Caucasian descent.

Alverine/simethicone is a combination of two drugs: Alverine citrate relaxes muscle cramps that occur in the intestine in conditions such as irritable bowel syndrome and diverticulosis. Simethicone is an antifoam administered orally. Reduces gas formation and facilitates its elimination from the digestive tract

ELIGIBILITY:
Inclusion Criteria:

* Subjects attending Hospital Juarez de Mexico with a diagnosis of diarrhea-predominant or mixed irritable bowel syndrome (IBS-D and IBS-M), according to Rome-IV criteria (Lacy et al. Gastroenterology 2016), providing Informed Consent.

Exclusion Criteria:

* Unexplained weight loss, blood in feces, anemia.
* Use of systemic antibiotics, NSAIDs, antipsychotic or prokinetic medication in the 3 weeks before study initiation.
* Pregnant or lactating women.
* History of gastrointestinal cancer.
* Suspicion of coeliac disease, inflammatory bowel disease (IBD), endometriosis or pelvic inflammatory disease.
* History of abdominal surgery within 2 years (3 months if appendectomy or herniorraphy)
* BMI below 18
* Known allergy to any of the components in the treatments

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-08-27 (Actual)

PRIMARY OUTCOMES:
Disease-specific quality of life (QoL) | 6 weeks
  Irritable bowel syndrome-specific validated IBSQoL questionnaire (Hahn et al. Aliment Pharmacol Ther 1997). Response is defined as an improvement of 15 or more points in the normalized 0-100 score

SECONDARY OUTCOMES:
Abdominal Pain | 6 weeks
  Abdominal Pain Visual Analog Scale, ranging 0 to 10 (i.e. 11-point scale, as recommended by FDA, May 2012 Guidance on Irritable Bowel Syndrome - Clinical Evaluation of Products for Treatment). Response is defined as an improvement of 30% at the end of the intervention compared to baseline.
Diarrhea | 6 weeks
  Stool consistency as determined with the Bristol scale (Lewis & Heaton, Scand. J. Gastroenterol 1997). Response is defined as a score equal or below 5 at the end of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Nuria Lopez Perez, MD, Study Director — Hospital Juarez de Mexico
Locations (1):
- Hospital Juarez de Mexico, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No